CLINICAL TRIAL: NCT06134674
Title: The Role of Early Enteral Nutrition in Critical Patients With COVID-19: A Retrospective Study
Brief Title: Early Versus Delayed Enteral Nutrition in Critically Ill Adults With COVID-19
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Selen Özsoy, Doctor of Philosophy, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCHBilkent-NUTR-EEN
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Enteral Nutrition; COVID-19 Acute Respiratory Distress Syndrome
Keywords: SARS-COV-2,COVID-19,intensive care unit,early enteral nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Enteral Nutrition: Patients who received enteral nutrition within the first 48 hours following intubation were included in the Early Enteral Nutrition (EEN) group.
- Late Enteral Nutrition: Patients who received enteral nutrition 48 hours or later following intubation were included in the late Enteral Nutrition (LEN) group.

SUMMARY:
The goal of this observational study is to determine the relationship between the nutritional profile of critically ill patients diagnosed with COVID-19 and disease severity, prognosis, and survival, to assess the ability to meet nutritional goals, EN complications, and reasons for discontinuation and postponement of feeding.

The main questions aim to answer are the relationship between the duration of EN initiation and Prognostic Nutritional Index (PNI) score, neutrophil-lymphocyte ratio (NLR), oxygenation status, MV, ICU, and length of hospital stay, overall mortality, and whether nutritional goals were met, EN complications, and reasons for discontinuation and postponement.

DETAILED DESCRIPTION:
Nutritional support is a crucial component of managing critically ill patients. The prognostic impact of early enteral nutrition (EN) in critically ill COVID-19 patients is largely unknown. The study aimed to determine the relationship between the nutritional profile of critically ill patients diagnosed with COVID-19 and disease severity, prognosis, and survival, to assess the ability to meet nutritional goals, EN complications, and reasons for discontinuation and postponement of feeding. Methods: This retrospective study was conducted with adult intensive care unit (ICU) patients diagnosed with COVID-19 and receiving mechanical ventilation (MV) and EN. The demographic, clinical, biochemical, and nutritional data of the patients were obtained from the patient's files and the hospital database. The initiation time, route, method, product type, amount, and duration of feeding were recorded, and the daily intake of energy, protein, pulp, and water were calculated. The nutritional requirements of the patients were defined, and achievement of targets, EN complications, and reasons for discontinuation and postponement were recorded. Patients were divided into two groups: early EN (EEN) if the feeding was initiated within the first 48 hours after MV and late EN (LEN) if 48 hours or later. The research outcomes are to determine the relationship between the duration of EN initiation and Prognostic Nutritional Index (PNI) score, neutrophil-lymphocyte ratio (NLR), oxygenation status, MV, ICU, and length of hospital stay, overall mortality, and whether nutritional goals were met, EN complications, and reasons for discontinuation and postponement.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with COVID-19
* aged 19 years and older
* on MV
* receiving only enteral tube nutrition

Exclusion Criteria:

* patients with an inflammatory disease
* myocardial infarction, collapse, and circulatory shock within the last 6 months
* hemodynamic instability
* embolism and stroke
* presence of unspecified coma
* renal disease
* cancer with a mortality rate of more than 50% within 6 months
* allogeneic bone marrow transplantation within 5 years
* enteral nutrition was contraindicated
* patients with allergic reactions to the enteral formula
* patients who received antioxidant supplements during feeding
* patients who received tube feeding supplemented with immunonutrition agents
* patients whose data could not be accurately retrieved

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study was conducted in a 3rd line ICU. The study included adult patients diagnosed with COVID-19, aged 19 years and older, on MV, and receiving enteral tube nutrition.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
mechanical ventilation (MV), intensive care unit (ICU), length of hospital stay and overall mortality. | through study completion, an average of 9 months
  The research outcomes are to determine the relationship between the duration of EN initiation and MV, ICU, and length of hospital stay, overall mortality.
Prognostic Nutritional Index (PNI) score, neutrophil-lymphocyte ratio (NLR), oxygenation status | From date of hospitalization and intubation until the date of extubation or date of death from any cause, whichever came first, assessed up to 9 months
  The research outcomes are to determine the relationship between the duration of EN initiation and Prognostic Nutritional Index (PNI) score, neutrophil-lymphocyte ratio (NLR), oxygenation status
Whether Nutritional goals were met, EN complications, and reasons for discontinuation and postponement. | From date of intubation until the date of extubation or date of death from any cause, whichever came first, assessed up to 9 months
  The research outcomes are to determine the relationship between the duration of EN initation and nutritional goals were met, EN complications, and reasons for discontinuation and postponement.

CONTACTS AND LOCATIONS:
Overall Officials: Selen Özsoy, PHD, Principal Investigator — Ankara City Hospital Bilkent; Mendane Saka, Prof.Dr., Study Director — Baskent University; Levent Öztürk, Prof.Dr., Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No